CLINICAL TRIAL: NCT01851616
Title: Oral Glucosestimulation After Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EKBB 298/12/1
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: glucose, blood
MeSH Terms: conditions — Obesity | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glucose 25g (Active Comparator): 25g of glucose in 200ml tap water, given orally (plus 50 mg 13C-sodium acetate)
  Interventions: Dietary Supplement: 25g of glucose in 200ml tap water, given orally (plus 50 mg 13C-sodium acetate)
- Glucose 10g (Active Comparator): 10g Glucose in 200ml tap water given orally (plus 50 mg 13C-sodium acetate)
  Interventions: Dietary Supplement: 10g Glucose in 200ml tap water given orally (plus 50 mg 13C-sodium acetate)

INTERVENTIONS:
Dietary Supplement: 25g of glucose in 200ml tap water, given orally (plus 50 mg 13C-sodium acetate)
  Arms: Glucose 25g
Dietary Supplement: 10g Glucose in 200ml tap water given orally (plus 50 mg 13C-sodium acetate)
  Arms: Glucose 10g

SUMMARY:
The objective of this study is to examine gastric emptying and satiety hormones after oral glucose stimulation in 2 different concentrations in morbidly obese patients after Roux-en-Y-gastric-Bypass.

DETAILED DESCRIPTION:
After gastric bypass many patients suffer from early and/or late dumping syndrome as a reaction to carbohydrate rich meals. Gastric emptying after bypass is accelerated and nutrition enters the intestine faster, which leads to osmotically driven fluid shifts from the blood to the lumen. Late dumping occurs 1-3 h after eating, and is caused by hyperinsulinemia and is therefore characterized by symptoms of hypoglycemia like weakness, sweating, and dizziness. Many people have both types. In most studies examining satiety hormones after oral glucose stimulation in non-operated patients, glucose loads of 50-75g are used. For a measurable GLP-1 rise a threshold of 2 kcal/min. at the intestine is needed. After gastric bypass gastric emptying is accelerated and less glucose is necessary to reach this threshold. The "threshold load" and "tolerable load without dumping symptoms" is not yet know.

ELIGIBILITY:
Inclusion Criteria:

* 6 weeks post gastric bypass surgery,
* non-diabetic patient

Exclusion Criteria:

* smoker,
* diabetes,
* gastrointestinal motility disorder,
* medication influencing gastric emptying

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
amount of oral glucose leading to increase in satiety hormones | 240 min.

SECONDARY OUTCOMES:
Amount of oral glucose leading to clinical signs of dumping | 240min.

OTHER OUTCOMES:
Gastric emptying after gastric bypass | 240min
  Gastric emptying is measured by means of breath test (use of 50 mg 13C-sodium acetate)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Prof., Principal Investigator — University of Basel
Locations (1):
- University Hospital of Basel, Basel, Switzerland